CLINICAL TRIAL: NCT07239999
Title: Randomized Controlled Trial Comparing Spinal Anesthesia With 1% Chloroprocaine Versus 1% Mepivacaine in Patients Undergoing Outpatient Primary Total Knee Arthroplasty
Brief Title: Comparing Spinal Anesthesia With 1% Chloroprocaine Versus 1% Mepivacaine in Patients Undergoing Outpatient Primary Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Husam Nashnoush, Doctor Husam Nashnoush, MBBCH, FRCPC, Anesthesia Department, Central Zone, DGH, Halifax , NS, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DGH2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Recovery Period; Anesthesia
Keywords: Spinal anesthesia; Outpatient total knee arthroplasty; Mepivacaine; Chloroprocaine
MeSH Terms: interventions — Mepivacaine; chloroprocaine

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Surgeons, PACU Nurses, OR Nurses, Physical therapists
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- One arm receives spinal Mepivacaine 50 mg (Active Comparator): One arm receives spinal Mepivacaine 50mg for total knee arthroplasty with adductor canal block
  Interventions: Drug: Mepivacaine Injection
- Spinal Chloroprocaine group (Active Comparator)
  Interventions: Drug: Chloroprocaine Injection

INTERVENTIONS:
Drug: Mepivacaine Injection — Comparing time to motor block recovery in PACU, time to PACU discharge, time to ambulation and length of hospital stay
  Arms: One arm receives spinal Mepivacaine 50 mg
Drug: Chloroprocaine Injection — Comparing time to motor block recovery in PACU, time to PACU discharge, time to ambulation and length of hospital stay
  Arms: Spinal Chloroprocaine group

SUMMARY:
This study or clinical trial looking to compare 2 types of freezing medications injected into the spinal fluid at the lower back between the vertebrae in patients going to have total knee replacement surgery to check for early legs movement, early discharge from recovery room, walking and hospital discharge. This could save hospital cost of such procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Elective outpatient TKA
* BMI less than 40
* Ability to provide surgical consent

Exclusion Criteria:

* Patient refusal
* Opioid tolerant
* Any contraindications to spinal anesthesia
* Chronic opioid use 3months or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-04-04 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Time to complete recovery of motor block | Time from the intrathecal drug injection to the first documented instance of complete motor block recovery Bromage 0. Within approximately 2 hours for the Chloroprocaine group and 4 hours for the Mepivacaine group.
Time to complete motor block recovery of lower limbs after spinal anesthesia | From the time of intrathecal drug injection to PACU discharge. Within approximately 3 hours for the Chloroprocaine group and 5 hours for the Mepivacaine group.
  Motor block will be assessed by PACU nurses in PACU using standard Bromage motor scale.

CONTACTS AND LOCATIONS:
Overall Officials: HUSAM M NASHNOUSH, MBBCH, FRCPC, Principal Investigator — Dalhousie University

IPD SHARING:
Plan to Share IPD: Yes
Patient data as Age, sex, BMI, drug doses, time to motor block, time to PACU discharge, time to ambulation, and LOS.
Supporting Information: Study Protocol
Time Frame: Jan2026 to Jan.2027
Access Criteria: Anesthesia Department, Dalhousie University Research Office
URL: https://clinicaltrials.gov

REFERENCES:
- [Background] Herndon CL, Martinez R, Sarpong NO, Geller JA, Shah RP, Cooper HJ. Spinal Anesthesia Using Chloroprocaine is Safe, Effective, and Facilitates Earlier Discharge in Selected Fast-track Total Hip Arthroplasty. Arthroplast Today. 2020 Jun 1;6(3):305-308. doi: 10.1016/j.artd.2020.04.007. eCollection 2020 Sep. PMID 32509943
- [Background] Callaghan JJ, Mont MA. Editorial: Proceedings of the Knee Society: A Knee Society-Journal of Arthroplasty Collaborative Partnership! J Arthroplasty. 2022 Jun;37(6S):S1. doi: 10.1016/j.arth.2022.02.078. Epub 2022 Feb 26. No abstract available. PMID 35227811
- [Background] Teunkens A, Vermeulen K, Van Gerven E, Fieuws S, Van de Velde M, Rex S. Comparison of 2-Chloroprocaine, Bupivacaine, and Lidocaine for Spinal Anesthesia in Patients Undergoing Knee Arthroscopy in an Outpatient Setting: A Double-Blind Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):576-83. doi: 10.1097/AAP.0000000000000420. PMID 27281722
- [Background] Lacasse MA, Roy JD, Forget J, Vandenbroucke F, Seal RF, Beaulieu D, McCormack M, Massicotte L. Comparison of bupivacaine and 2-chloroprocaine for spinal anesthesia for outpatient surgery: a double-blind randomized trial. Can J Anaesth. 2011 Apr;58(4):384-91. doi: 10.1007/s12630-010-9450-x. Epub 2011 Jan 4. PMID 21203878
- [Background] Gilreath N, Liu J, Thomson C, Daher M, Caus S, Dunn H, Antoci V Jr, Barrett T, Cohen E. Retrospective comparison of chloroprocaine and mepivacaine in spinal anesthesia for same-day discharge TKA. Knee Surg Relat Res. 2025 Aug 7;37(1):33. doi: 10.1186/s43019-025-00283-4. PMID 40775385
- [Background] Alhefeiti K, Patrascu AM, Lustig S, Aubrun F, Dziadzko M. Perioperative Outcomes in Patients Who Received Spinal Chloroprocaine for Total Hip or Knee Arthroplasty-Consecutive Case Series Study. J Clin Med. 2022 Sep 29;11(19):5771. doi: 10.3390/jcm11195771. PMID 36233638
- [Background] Ghisi D, Boschetto G, Spinelli AM, Giannone S, Frugiuele J, Ciccarello M, Bonarelli S. Spinal anaesthesia with Chloroprocaine HCl 1% for elective lower limb procedures of short duration: a prospective, randomised, observer-blind study in adult patients. BMC Anesthesiol. 2021 Feb 20;21(1):58. doi: 10.1186/s12871-021-01279-9. PMID 33610175
- [Background] Pillow CF, Brewbaker C, Wolf BJ, Barrett W, Hansen E, Brown A, Crawford D, Wilson SH. Mepivacaine versus bupivacaine spinal anesthesia for return of motor function following total knee arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2025 May 1:rapm-2024-106342. doi: 10.1136/rapm-2024-106342. Online ahead of print. PMID 40316299
- [Background] Schwenk ES, Kasper VP, Smoker JD, Mendelson AM, Austin MS, Brown SA, Hozack WJ, Cohen AJ, Li JJ, Wahal CS, Baratta JL, Torjman MC, Nemeth AC, Czerwinski EE. Mepivacaine versus Bupivacaine Spinal Anesthesia for Early Postoperative Ambulation. Anesthesiology. 2020 Oct 1;133(4):801-811. doi: 10.1097/ALN.0000000000003480. PMID 32852904
- [Background] Forster JG. Short-acting spinal anesthesia in the ambulatory setting. Curr Opin Anaesthesiol. 2014 Dec;27(6):597-604. doi: 10.1097/ACO.0000000000000126. PMID 25211156
- [Background] Siddiqi A, Mahmoud Y, Secic M, Tozzi JM, Emara A, Piuzzi NS, Culp B, Schwarzkopf R, Springer BD, Chen AF. Mepivacaine Versus Bupivacaine Spinal Anesthesia for Primary Total Joint Arthroplasty: A Systematic Review and Meta-Analysis. J Arthroplasty. 2022 Jul;37(7):1396-1404.e5. doi: 10.1016/j.arth.2022.03.031. Epub 2022 Mar 17. PMID 35306162
- [Background] Wyles CC, Pagnano MW, Trousdale RT, Sierra RJ, Taunton MJ, Perry KI, Larson DR, Amundson AW, Smith HM, Duncan CM, Abdel MP. More Predictable Return of Motor Function with Mepivacaine Versus Bupivacaine Spinal Anesthetic in Total Hip and Total Knee Arthroplasty: A Double-Blinded, Randomized Clinical Trial. J Bone Joint Surg Am. 2020 Sep 16;102(18):1609-1615. doi: 10.2106/JBJS.20.00231. PMID 32960532
- [Background] Mahan MC, Jildeh TR, Tenbrunsel TN, Davis JJ. Mepivacaine Spinal Anesthesia Facilitates Rapid Recovery in Total Knee Arthroplasty Compared to Bupivacaine. J Arthroplasty. 2018 Jun;33(6):1699-1704. doi: 10.1016/j.arth.2018.01.009. Epub 2018 Jan 16. PMID 29429882
- [Background] Camponovo C, Wulf H, Ghisi D, Fanelli A, Riva T, Cristina D, Vassiliou T, Leschka K, Fanelli G. Intrathecal 1% 2-chloroprocaine vs. 0.5% bupivacaine in ambulatory surgery: a prospective, observer-blinded, randomised, controlled trial. Acta Anaesthesiol Scand. 2014 May;58(5):560-6. doi: 10.1111/aas.12291. Epub 2014 Mar 6. PMID 24601887
- [Background] Casati A, Fanelli G, Danelli G, Berti M, Ghisi D, Brivio M, Putzu M, Barbagallo A. Spinal anesthesia with lidocaine or preservative-free 2-chlorprocaine for outpatient knee arthroscopy: a prospective, randomized, double-blind comparison. Anesth Analg. 2007 Apr;104(4):959-64. doi: 10.1213/01.ane.0000258766.73612.d8. PMID 17377114
- [Background] Goldblum E, Atchabahian A. The use of 2-chloroprocaine for spinal anaesthesia. Acta Anaesthesiol Scand. 2013 May;57(5):545-52. doi: 10.1111/aas.12071. Epub 2013 Jan 16. PMID 23320599
- [Background] Capdevila X, Aveline C, Delaunay L, Bouaziz H, Zetlaoui P, Choquet O, Jouffroy L, Herman-Demars H, Bonnet F. Impact of Chloroprocaine on the Eligibility for Hospital Discharge in Patients Requiring Ambulatory Surgery Under Spinal Anesthesia: An Observational Multicenter Prospective Study. Adv Ther. 2020 Jan;37(1):541-551. doi: 10.1007/s12325-019-01172-5. Epub 2019 Dec 11. PMID 31828611
- [Background] Wesselink E, Hurk GJD, Vegt RV, Slagt C, Aa JV, Franssen E, Ven PV, Swart N, Boer C, Leeuw M. Chloroprocaine versus prilocaine for spinal anesthesia in ambulatory knee arthroscopy: a double-blind randomized trial. Reg Anesth Pain Med. 2019 Aug 21:rapm-2019-100673. doi: 10.1136/rapm-2019-100673. Online ahead of print. PMID 31439640
- [Background] Kim SW, Khandaker R, Muse IO, Pulverenti T, Goman M, Patel J, Yedlin A, Balikai CP, Levine R, Choice C, Montilla Medrano E. Comparison of 1% chloroprocaine hydrochloride versus hyperbaric bupivacaine spinal in patients undergoing anorectal surgery in an ambulatory surgery center: a double-blind randomized clinical trial. Reg Anesth Pain Med. 2024 Dec 31:rapm-2024-106130. doi: 10.1136/rapm-2024-106130. Online ahead of print. PMID 39740957
- [Background] Singh NP, Siddiqui NT, Makkar JK, Guffey R, Singh PM. Optimal local anesthetic for spinal anesthesia in patients undergoing ambulatory non-arthroplasty surgery: a systematic review and Bayesian network meta-analysis of randomized controlled trials. Can J Anaesth. 2025 Apr;72(4):550-566. doi: 10.1007/s12630-025-02924-4. Epub 2025 Apr 8. PMID 40199797
- [Background] Forget P, Borovac JA, Thackeray EM, Pace NL. Transient neurological symptoms (TNS) following spinal anaesthesia with lidocaine versus other local anaesthetics in adult surgical patients: a network meta-analysis. Cochrane Database Syst Rev. 2019 Dec 1;12(12):CD003006. doi: 10.1002/14651858.CD003006.pub4. PMID 31786810
- [Background] Khurana BJK, Choudhary S, Singhal M, Rautela RS, Salhotra R, Singh A, Meena S. Comparison of Intrathecal Chloroprocaine With Bupivacaine in Short Gynecological Procedures: A Randomized Double-Blind Study. Cureus. 2023 Aug 27;15(8):e44187. doi: 10.7759/cureus.44187. eCollection 2023 Aug. PMID 37767250
- [Background] Gu L, Smith CR, Ihnatsenka B, Zasimovich Y, Le-Wendling L. Comparing Spinal Chloroprocaine to Hyperbaric and Isobaric Bupivacaine for Total Hip and Knee Arthroplasties: A Retrospective Study. Cureus. 2023 Mar 3;15(3):e35729. doi: 10.7759/cureus.35729. eCollection 2023 Mar. PMID 37016653